CLINICAL TRIAL: NCT01950130
Title: Prophylactic Preoperative Inatraaortic Balloon Pump (IABP) in High-risk Patients Undergoing Coronary Artery Bypass Surgery (CABG)
Brief Title: Prophylactic IABP in High-risk Patients Undergoing CABG
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding
Sponsor: University of Giessen (Other)
Responsible Party: Principal Investigator, Dr. Philippe Grieshaber, MD, University of Giessen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-1124
Record Dates: First submitted 2013-09-18; First posted 2013-09-25 (Estimated); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Myocardial Infarction; Coronary Artery Disease
Keywords: IABP; IABC; coronary artery disease; prophylactic; cardiac assist
MeSH Terms: conditions — Myocardial Infarction; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IABP group (Experimental): Preoperative IABP insertion
  Interventions: Procedure: Preoperative IABC
- Control group (No Intervention): Preoperative conservative treatment

INTERVENTIONS:
Procedure: Preoperative IABC — IABP-Insertion upon inclusion into the trial and admission to the ICU
  Arms: IABP group

SUMMARY:
Due to advances and increased practice of interventional therapy for coronary artery disease, the rate of high-risk patients with severe coronary disease and reduced left ventricular function among patients undergoing coronary artery bypass grafting surgery (CABG) is increasing. The perioperative mortality in these patients is ≥ 5%. The perioperative and operative management for these patients has to be optimized in order to reduce their perioperative morbidity and mortality. One of the central aspects is perioperative maintenance of hemodynamic stability. The use of prophylactic IABP is a partly established, but not sufficiently evidence-based measure to reduce ventricular afterload and improve coronary perfusion pre-, intra- and postoperatively. Yet, it is an invasive procedure with potential complications. The planned trial should give an explicit answer, whether preoperative prophylactic IABP decreases 30-day all-cause mortality (primary endpoint) and long-term mortality (3, 6, 12 months; secondary endpoints) compared to preoperative conservative treatment in high-risk patients undergoing CABG.

ELIGIBILITY:
Key inclusion criteria:

Hemodynamically stable high-risk patients before CABG, defined by the following criteria:

* Age >18 years
* Isolated CABG planned
* Informed consent in trial participation given
* Any left ventricular functional impairment (regional wall motion abnormality or global LVEF<55%) assessed via ventriculography or transthoracic or transeophageal echocardiography
* Elevated cardiac biomarkers (CK-MB > 6% of total-CK, Troponin I > 3-fold of specific test reference) or myocardial infarction (NSTEMI or STEMI) within the last 4 days.

Key exclusion criteria:

* Contraindications for IABP
* Cardiogenic shock
* Shock of any other cause
* Critical preoperative state according to EuroSCORE II-criteria
* Cardiac surgical procedure other than CABG planned
* Severe comorbidity with life expectancy < 6 months
* Incapability of giving informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2017-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
30-day all-cause mortality post CABG [%] | 30 days

SECONDARY OUTCOMES:
Survival at 3, 6, 12 months [%] | 3, 6 and 12 months
Duration of ICU stay [h] | 48 hours (average)
Dependence on medical inotropic support | 48 hours (average)
IABP-associated complications | 8 days (average)
  IABP-associated complications occur most often during IABP-support. However, after weaning from IABP, patients can still have bleeding complications or thrombembolic complications. Therefore, IABP-associated complications are monitored during the whole hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Grieshaber, MD, Study Director — Giessen University
Locations (1):
- Department of Adult and Pediatric Cardiovascular Surgery, Giessen, Germany